CLINICAL TRIAL: NCT06489353
Title: The Effect of Watching Video and Blowing Paper Pinwheels on Pain and Fear in Children Undergoing Venipuncture.
Brief Title: The Effect of Watching Video and Blowing Paper Pinwheels in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, HuiMing Hou, Head Nurse, Department of Nursing, Taichung Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CF24157B
Record Dates: First submitted 2024-06-05; First posted 2024-07-05 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Pain; Fear
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Participants will:
  * Be randomly assigned to one of three groups in parallel for the duration of the study:
  * Watch their preferred cartoons on an iPad during the venipuncture process.
  * Blow paper pinwheels to distract themselves during the venipuncture process.
  * Receive standard care without any additional distractions.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: 1. Randomization and Allocation: Participants are randomly assigned to one of three groups using a computer-generated table. Group assignments are sealed in opaque envelopes and revealed by a research coordinator not involved in assessments.
  2. Blinding Care Providers: The nurse is unaware of the group assignment. The coordinator informs the parent and child of the intervention just before the procedure.
  3. Blinding outcomes assessor: Outcome assessors and data analysts are kept blind to group assignments and only receive anonymized data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Video-watching group (Experimental): Participants will watch age-appropriate and engaging videos during the venipuncture procedure to distract them from pain and fear.
  Interventions: Behavioral: Video-watching
- Blowing Pinwheels (Experimental): Participants will blow pinwheels during the venipuncture procedure, using breathing control and distraction to reduce pain and fear.
  Interventions: Behavioral: Blowing Pinwheels
- routine care group (No Intervention): Participants will receive standard routine care during the venipuncture procedure without additional interventions, serving as the control group.

INTERVENTIONS:
Behavioral: Video-watching — Participants will watch age-appropriate and engaging videos.
  Arms: Video-watching group
Behavioral: Blowing Pinwheels — Participants will blow pinwheels during the venipuncture procedure
  Arms: Blowing Pinwheels

SUMMARY:
The goal of this clinical trial is to evaluate if watching videos and blowing paper pinwheels can reduce pain and fear in children undergoing venipuncture. The participant population includes hospitalized children aged 3-6 years old undergoing venipuncture for the first time.

The main questions it aims to answer are:

1. Does watching videos reduce pain and fear during venipuncture in children?
2. Does blowing paper pinwheels reduce pain and fear during venipuncture in children?

Researchers will compare a group watching videos and a group blowing paper pinwheels to a control group receiving standard care to see if these interventions reduce pain and fear.

Participants will:

* Watch their preferred cartoons on an iPad during the venipuncture process.
* Blow paper pinwheels to distract themselves during the venipuncture process.
* Be accompanied by a family member who will help in holding the child and providing comfort.

DETAILED DESCRIPTION:
The goal of this clinical trial is to explore the effectiveness of watching videos and blowing paper pinwheels in reducing pain and fear in children undergoing venipuncture in children aged 3-6 years hospitalized for the first time and undergoing intravenous infusion or blood draw. The main questions it aims to answer are:

* Does watching videos reduce the pain experienced by children during venipuncture?
* Does blowing paper pinwheels reduce the fear experienced by children during venipuncture?

If there is a comparison group: Researchers will compare the group of children watching videos and the group of children blowing paper pinwheels to the control group receiving standard care to see if these interventions are effective in reducing pain and fear during venipuncture.

Participants will:

* Be children aged 3-6 years hospitalized for the first time and undergoing intravenous infusion or blood draw.
* Have no chronic diseases, developmental delays, or epilepsy.
* Have no difficulty speaking, auditory or visual impairments, and have not used sedatives within 6 hours prior to the procedure.

Interventions:

Participants will be randomly assigned to one of three groups:

1. Video Watching Group:

   * Children will choose their preferred cartoon videos.
   * They will watch the video on an iPad for 1 minute before and during venipuncture.
   * Parents will assist in stabilizing the child and providing comfort during the procedure.
2. Paper Pinwheel Blowing Group:

   * Children will select a paper pinwheel of their choice.
   * They will practice blowing the pinwheel for 1 minute before the procedure.
   * During venipuncture, they will blow the pinwheel with parental assistance for stabilization and comfort.
3. Control Group:

   * Children will receive standard care with parental presence but no additional interventions during venipuncture.
   * After the procedure, children will be allowed to play a "pinprick" game and choose a small toy as a reward.

Outcome Measures

The effectiveness of the interventions will be measured using the following tools

1. The Wong-Baker Faces Pain Scale (WBFPS):

   * Used to assess children's self-reported pain levels before and after venipuncture.
   * Scores range from 0 to 10, with higher scores indicating greater pain.
2. Parental State Anxiety Scale:

   * A Chinese version of the state anxiety scale will be used to measure parents' anxiety levels.
   * Scores range from 1 to 4 for each item, with higher scores indicating greater anxiety.
3. Parental Satisfaction Scale:

   * A 0-10 scale will be used to measure parents' satisfaction with the venipuncture process.
4. The Children's Fear Scale:

   * Used to assess children's fear levels before and after venipuncture.
   * Scores range from 0 to 4, with higher scores indicating greater fear.
5. FLACC (Face, Legs, Activity, Cry, Consolability) Pain Assessment Scale:

   * Used to assess pain in non-verbal children based on facial expressions, leg movements, activity, cry, and consolability.
   * Scores range from 0 to 10, with higher scores indicating greater pain.

Study Design

This study will be conducted at the 66th Ward of Taichung Veterans General Hospital. After obtaining informed consent from parents and assent from children, participants will be randomly assigned to one of the three groups using a random number generator. The nurse performing the venipuncture will be blinded to the group assignment. Data will be collected by research personnel not involved in the data collection process.

Statistical Analysis

Descriptive statistics will include frequencies, means, and standard deviations. Inferential statistics will be conducted using ANOVA to determine the significance of the differences between groups.

Expected Outcomes

The study expects that children in the intervention groups (video watching and paper pinwheel blowing) will have lower pain and fear scores, and their parents will have lower anxiety scores and higher satisfaction compared to the control group. This research aims to improve the quality of care for hospitalized children undergoing venipuncture.

Handling of Adverse Reactions

If participants experience dizziness or discomfort during the intervention, the procedure will be stopped immediately, and necessary assistance will be provided.

Funding and Compensation

The study is funded by the Taichung Veterans General Hospital internal research project (project number: TCVGH-1137404B). Any adverse reactions caused by the study will be covered by the hospital, excluding anticipated side effects listed in the informed consent form.

Conflict of Interest There are no potential conflicts of interest associated with this study.

ELIGIBILITY:
Inclusion Criteria:

* aged 3-6 years.
* undergoing intravenous infusion or blood draw during the hospital stay.

Exclusion Criteria:

* chronic diseases.
* developmental delays or epilepsy.
* difficulty speaking.
* hearing or visual impairments.
* use sedatives within the past 6 hours.
* history of fainting during intravenous infusion or blood draw.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 93 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2025-05-16 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Wong-Baker Faces Pain Scale (WBFPS) for Children's Self-Reported Pain | Assessed immediately before and after the venipuncture.
  The Wong-Baker Faces Pain Scale (WBFPS) is used to measure children's self-reported pain levels. It consists of a series of facial expressions ranging from a smiling face (0) indicating "no pain" to a crying face (10) indicating "worst pain." The child points to the face that best describes their pain.
FLACC (Face, Legs, Activity, Cry, Consolability) Behavioral Pain Assessment Scale | Assessed immediately before and after the venipuncture procedure.
  The FLACC scale is used to measure pain in children by evaluating five criteria: Face (facial expressions), Legs (movement and positioning), Activity (overall movement and muscle tone), Cry (verbal expressions of pain), and Consolability (the child's ability to be comforted). Each criterion is scored from 0 to 2, with a total score ranging from 0 to 10. Higher scores indicate greater pain severity.
Children's Fear Scale (CFS) | Assessed immediately before and after the venipuncture procedure.
  The Children's Fear Scale (CFS) is used to evaluate the level of fear experienced by children during venipuncture. The scale consists of five facial expressions ranging from a neutral face (0) indicating "no fear" to a very frightened face (4) indicating "high fear." The nurse observes the child's facial expressions and assigns a score based on the child's appearance and behavior during the procedure.

SECONDARY OUTCOMES:
Parental State Anxiety Scale (PSAS) | Assessed immediately after the child's venipuncture procedure.
  The Parental State Anxiety Scale (PSAS) measures the anxiety levels of parents during their child's venipuncture procedure. The scale consists of 20 items, with each item rated on a 4-point scale ranging from 1 (not at all) to 4 (very much). The total score ranges from 20 to 80, with higher scores indicating greater levels of anxiety. The scale assesses the parents' feelings of tension, nervousness, and worry in the specific context of their child's medical procedure.
Satisfaction of parents | Assessed immediately after the child's venipuncture procedure.
  A 0-10 scale is used to measure family members' satisfaction with the venipuncture process. After the venipuncture procedure, family members fill out this scale, with higher scores indicating greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Ming Hou, MD, Principal Investigator — Taichung Veterans' General Hospital
Locations (1):
- Taichung Veterans' General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shen T, Wang X, Xue Q, Chen D. Active versus passive distraction for reducing procedural pain and anxiety in children: a meta-analysis and systematic review. Ital J Pediatr. 2023 Aug 31;49(1):109. doi: 10.1186/s13052-023-01518-4. PMID 37653423
- [Background] Aydin D, Sahiner NC, Ciftci EK. Comparison of the effectiveness of three different methods in decreasing pain during venipuncture in children: ball squeezing, balloon inflating and distraction cards. J Clin Nurs. 2016 Aug;25(15-16):2328-35. doi: 10.1111/jocn.13321. Epub 2016 Apr 26. PMID 27112434
- [Background] Baxter AL, Cohen LL, McElvery HL, Lawson ML, von Baeyer CL. An integration of vibration and cold relieves venipuncture pain in a pediatric emergency department. Pediatr Emerg Care. 2011 Dec;27(12):1151-6. doi: 10.1097/PEC.0b013e318237ace4. PMID 22134226
- [Background] Hartling L, Newton AS, Liang Y, Jou H, Hewson K, Klassen TP, Curtis S. Music to reduce pain and distress in the pediatric emergency department: a randomized clinical trial. JAMA Pediatr. 2013 Sep;167(9):826-35. doi: 10.1001/jamapediatrics.2013.200. PMID 23857075
- [Background] Vetri Buratti C, Angelino F, Sansoni J, Fabriani L, Mauro L, Latina R. Distraction as a technique to control pain in pediatric patients during venipuncture. A narrative review of literature. Prof Inferm. 2015 Jan-Mar;68(1):52-62. doi: 10.7429/pi.2015.681052. PMID 25837616
- [Background] da Silva JR, Pizzoli LM, Amorim AR, Pinheiros FT, Romanini GC, da Silva JG, Joanete S, Alves SS. Using Therapeutic Toys to Facilitate Venipuncture Procedure in Preschool Children. Pediatr Nurs. 2016 Mar-Apr;42(2):61-8. PMID 27254974
- [Background] Rimon A, Shalom S, Wolyniez I, Gruber A, Schachter-Davidov A, Glatstein M. Medical Clowns and Cortisol levels in Children Undergoing Venipuncture in the Emergency Department: A Pilot Study. Isr Med Assoc J. 2016 Nov;18(11):680-683. PMID 28466619
- [Background] Piskorz J, Czub M. Effectiveness of a virtual reality intervention to minimize pediatric stress and pain intensity during venipuncture. J Spec Pediatr Nurs. 2018 Jan;23(1). doi: 10.1111/jspn.12201. Epub 2017 Nov 20. PMID 29155488
- [Background] Ballard A, Khadra C, Adler S, Doyon-Trottier E, Le May S. Efficacy of the Buzzy(R) device for pain management of children during needle-related procedures: a systematic review protocol. Syst Rev. 2018 May 22;7(1):78. doi: 10.1186/s13643-018-0738-1. PMID 29788987
- [Background] Susam V, Friedel M, Basile P, Ferri P, Bonetti L. Efficacy of the Buzzy System for pain relief during venipuncture in children: a randomized controlled trial. Acta Biomed. 2018 Jul 18;89(6-S):6-16. doi: 10.23750/abm.v89i6-S.7378. PMID 30038198
- [Background] Birnie KA, Noel M, Chambers CT, Uman LS, Parker JA. Psychological interventions for needle-related procedural pain and distress in children and adolescents. Cochrane Database Syst Rev. 2018 Oct 4;10(10):CD005179. doi: 10.1002/14651858.CD005179.pub4. PMID 30284240
- [Background] Chan E, Hovenden M, Ramage E, Ling N, Pham JH, Rahim A, Lam C, Liu L, Foster S, Sambell R, Jeyachanthiran K, Crock C, Stock A, Hopper SM, Cohen S, Davidson A, Plummer K, Mills E, Craig SS, Deng G, Leong P. Virtual Reality for Pediatric Needle Procedural Pain: Two Randomized Clinical Trials. J Pediatr. 2019 Jun;209:160-167.e4. doi: 10.1016/j.jpeds.2019.02.034. Epub 2019 Apr 29. PMID 31047650
- [Background] Dumoulin S, Bouchard S, Ellis J, Lavoie KL, Vezina MP, Charbonneau P, Tardif J, Hajjar A. A Randomized Controlled Trial on the Use of Virtual Reality for Needle-Related Procedures in Children and Adolescents in the Emergency Department. Games Health J. 2019 Aug;8(4):285-293. doi: 10.1089/g4h.2018.0111. Epub 2019 May 24. PMID 31135178
- [Background] Celikol S, Tural Buyuk E, Yildizlar O. Children's Pain, Fear, and Anxiety During Invasive Procedures. Nurs Sci Q. 2019 Jul;32(3):226-232. doi: 10.1177/0894318419845391. PMID 31203776
- [Background] Wong CL, Lui MMW, Choi KC. Effects of immersive virtual reality intervention on pain and anxiety among pediatric patients undergoing venipuncture: a study protocol for a randomized controlled trial. Trials. 2019 Jun 20;20(1):369. doi: 10.1186/s13063-019-3443-z. PMID 31221208
- [Background] Yilmaz Kurt F, Aytekin Ozdemir A, Atay S. The Effects of Two Methods on Venipuncture Pain in Children: Procedural Restraint and Cognitive-Behavioral Intervention Package. Pain Manag Nurs. 2020 Dec;21(6):594-600. doi: 10.1016/j.pmn.2019.09.002. Epub 2019 Oct 15. PMID 31628067
- [Background] Padoan A, Sirini S, Mazzone R, Mesiti C, Grillo C, Meyer B, Plebani M. Evaluation of an improved small gauge needle for venipuncture in children with difficult venous access: Impact on sample quality, phlebotomist satisfaction and patient pain perception. Clin Chim Acta. 2020 Jan;500:213-219. doi: 10.1016/j.cca.2019.10.019. Epub 2019 Oct 31. PMID 31678576
- [Background] Ozalp Gerceker G, Ayar D, Ozdemir EZ, Bektas M. Effects of virtual reality on pain, fear and anxiety during blood draw in children aged 5-12 years old: A randomised controlled study. J Clin Nurs. 2020 Apr;29(7-8):1151-1161. doi: 10.1111/jocn.15173. Epub 2020 Jan 22. PMID 31889358
- [Background] Arikan A, Esenay FI. Active and Passive Distraction Interventions in a Pediatric Emergency Department to Reduce the Pain and Anxiety During Venous Blood Sampling: A Randomized Clinical Trial. J Emerg Nurs. 2020 Nov;46(6):779-790. doi: 10.1016/j.jen.2020.05.004. Epub 2020 Jul 22. PMID 32711948
- [Background] Tibaldo C, Castagno E, Aguzzi S, Urbino AF. [Non pharmacologic interventions for pain associated to venipuncture in children: a literature review]. Assist Inferm Ric. 2020 Oct-Dec;39(4):179-187. doi: 10.1702/3508.34951. Italian. PMID 33362188
- [Background] Grabinski ZG, Boscamp NS, Zuckerman WA, Zviti R, O'Brien A, Martinez M, Tsze DS. Efficacy of Distraction for Reducing Pain and Distress Associated With Venipuncture in the Pediatric Posttransplant Population: A Randomized Controlled Trial. Pediatr Emerg Care. 2022 Feb 1;38(2):e811-e815. doi: 10.1097/PEC.0000000000002458. PMID 34034337
- [Background] Canares T, Parrish C, Santos C, Badawi A, Stewart A, Kleinman K, Psoter K, McGuire J. Pediatric Coping During Venipuncture With Virtual Reality: Pilot Randomized Controlled Trial. JMIR Pediatr Parent. 2021 Jul 28;4(3):e26040. doi: 10.2196/26040. PMID 34319249
- [Background] Sajeev MF, Kelada L, Yahya Nur AB, Wakefield CE, Wewege MA, Karpelowsky J, Akimana B, Darlington AS, Signorelli C. Interactive video games to reduce paediatric procedural pain and anxiety: a systematic review and meta-analysis. Br J Anaesth. 2021 Oct;127(4):608-619. doi: 10.1016/j.bja.2021.06.039. Epub 2021 Jul 31. PMID 34340838
- [Background] Lee HN, Bae W, Park JW, Jung JY, Hwang S, Kim DK, Kwak YH. Virtual reality environment using a dome screen for procedural pain in young children during intravenous placement: A pilot randomized controlled trial. PLoS One. 2021 Aug 31;16(8):e0256489. doi: 10.1371/journal.pone.0256489. eCollection 2021. PMID 34464411
- [Background] Fusetti V, Re L, Pigni A, Tallarita A, Cilluffo S, Caraceni AT, Lusignani M. Clown therapy for procedural pain in children: a systematic review and meta-analysis. Eur J Pediatr. 2022 Jun;181(6):2215-2225. doi: 10.1007/s00431-022-04440-9. Epub 2022 Mar 16. PMID 35294645
- [Background] Ali S, Rajagopal M, Stinson J, Ma K, Vandermeer B, Felkar B, Schreiner K, Proctor A, Plume J, Hartling L. Virtual reality-based distraction for intravenous insertion-related distress in children: a study protocol for a randomised controlled trial. BMJ Open. 2022 Mar 30;12(3):e057892. doi: 10.1136/bmjopen-2021-057892. PMID 35354617
- [Background] Ugucu G, Akdeniz Uysal D, Guzel Polat O, Artuvan Z, Polat Kulcu D, Aksu D, Gulgun Altintas M, Cetin H, Orekici Temel G. Effects of cartoon watching and bubble-blowing during venipuncture on pain, fear, and anxiety in children aged 6-8 years: A randomized experimental study. J Pediatr Nurs. 2022 Jul-Aug;65:e107-e114. doi: 10.1016/j.pedn.2022.03.016. Epub 2022 Apr 8. PMID 35410736
- [Background] Ryu JH, Han SH, Hwang SM, Lee J, Do SH, Kim JH, Park JW. Effects of Virtual Reality Education on Procedural Pain and Anxiety During Venipuncture in Children: A Randomized Clinical Trial. Front Med (Lausanne). 2022 Apr 7;9:849541. doi: 10.3389/fmed.2022.849541. eCollection 2022. PMID 35463010
- [Background] Suleman SK, Atrushi A, Enskar K. Effectiveness of art-based distraction on reducing pediatric patients' pain and anxiety during venipuncture: A randomized controlled trial. Complement Ther Clin Pract. 2022 Aug;48:101597. doi: 10.1016/j.ctcp.2022.101597. Epub 2022 Apr 30. PMID 35512482
- [Background] Azak M, Aksucu G, Caglar S. The Effect of Parental Presence on Pain Levels of Children During Invasive Procedures: A Systematic Review. Pain Manag Nurs. 2022 Oct;23(5):682-688. doi: 10.1016/j.pmn.2022.03.011. Epub 2022 May 4. PMID 35523626
- [Background] Constantin KL, Moline RL, Pillai Riddell R, Spence JR, Fiacconi CM, Lupo-Flewelling K, McMurtry CM. Parent and child self- and co-regulation during pediatric venipuncture: Exploring heart rate variability and the effects of a mindfulness intervention. Dev Psychobiol. 2022 Jul;64(5):e22277. doi: 10.1002/dev.22277. PMID 35603416
- [Background] Semerci R, Akarsu O, Kilic D. The effect of buzzy and cold spray on pain, anxiety, and fear of children during venipuncture in pediatric emergency department in Turkey; A randomized controlled study. J Pediatr Nurs. 2023 Jan-Feb;68:e1-e7. doi: 10.1016/j.pedn.2022.08.019. Epub 2022 Sep 9. PMID 36089558
- [Background] Halal Mehdi Alfatavi H, Sadeghi T, Baqer Hassan Mohammed Al-Dakheel M, Asadi Noghabi F, Sahebkar Moeini M. Effects of Whistling Compared with Buzzy Device During Blood Sampling on Pain and Fear in Children's Emergency Department. Compr Child Adolesc Nurs. 2022 Dec;45(4):414-424. doi: 10.1080/24694193.2022.2091683. Epub 2022 Jul 11. PMID 36440867
- [Background] Yu Z, Zhou Y, Xu X, Lin L, Le Q, Gu Y. Pharmacological and non-pharmacological interventions in management of peripheral venipuncture-related pain: a randomized clinical trial. BMC Pediatr. 2023 Feb 3;23(1):58. doi: 10.1186/s12887-023-03855-z. PMID 36737707
- [Background] Wong CL, Choi KC. Effects of an Immersive Virtual Reality Intervention on Pain and Anxiety Among Pediatric Patients Undergoing Venipuncture: A Randomized Clinical Trial. JAMA Netw Open. 2023 Feb 1;6(2):e230001. doi: 10.1001/jamanetworkopen.2023.0001. PMID 36795410